CLINICAL TRIAL: NCT04185792
Title: Polish Translation and Validation of the Neurogenic Bladder Symptom Score (NBSS), Qualiveen and Short Form Qualiveen (SF-Qualiveen) Questionnaires
Brief Title: Polish Translation and Validation of NBSS, Qualiveen and SF-Qualiveen
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Collaborators: Piotr Chlosta, Full-time Professor, University Hospital, Cracow, Poland (Unknown)
Responsible Party: Principal Investigator, Mikolaj Przydacz, Assistant Professor, Principal Investigator, Jagiellonian University
Other Study IDs: 1072.6120.222.2019
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Spinal Cord Injuries; Multiple Sclerosis
MeSH Terms: conditions — Spinal Cord Injuries; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with spinal cord injury: NBSS, Qualiveen and SF-Qualiveen questionnaires will be administered to participants.
  Interventions: Diagnostic Test: NBSS, Qualiveen and SF-Qualiveen
- Patients with multiple sclerosis: NBSS, Qualiveen and SF-Qualiveen questionnaires will be administered to participants.
  Interventions: Diagnostic Test: NBSS, Qualiveen and SF-Qualiveen

INTERVENTIONS:
Diagnostic Test: NBSS, Qualiveen and SF-Qualiveen — NBSS, Qualiveen and SF-Qualiveen are self-reported questionnaires.

SUMMARY:
The aim of this study is to translate, culturally adapt, and validate Polish versions of the NBSS, Qualiveen and SF-Qualiveen questionnaires.

DETAILED DESCRIPTION:
The aim of this study is to translate, culturally adapt, and validate Polish versions of the NBSS, Qualiveen and SF-Qualiveen questionnaires in patients with spinal cord injury and multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury patients
* Multiple sclerosis patients
* Age > 18

Exclusion Criteria:

* Spinal shock patients
* Urinary tract operation in the last month
* Quality of life changes in the last month
* Urinary tract infections in the last month
* Bladder management changes or drug changes in the last month

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 200 patients with spinal cord injury and multiple sclerosis
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
ICIQ-SF | 6 months
  The ICIQ-SF questionnaire is a brief questionnaire that was devised to assess the burden of urinary incontinence in a patient's life, evaluating its impact on patients' QoL. It is composed by four questions that evaluate frequency, severity, and impact of incontinence on QoL and another section evaluating usual urinary loss situations. The minimum and maximum values range between 0-21 points. Higher the score, the greater the severity of the symptoms.
  The ICIQ-SF has been chosen as the validation questionnaire.
Neurogenic Bladder Symptom Score Questionnaire (NBSS) | 6 months
  Neurogenic Bladder Symptom Score Questionnaire is a 24 item self-reported questionnaire (0-74 points). The questionnaire includes 4 subgroups; incontinence (0-29 points), storage&voiding (0-22 points) and consequences (0-23 points). Higher the score, the greater the severity of the symptoms.
Qualiveen | 6 months
  The Qualiveen is divided in two major sections-Specific Impact of Urinary Problems on Quality of Life (SIUP) and General Quality of Life (GQoL).
  The first part, specific for urinary problems, has a total of 30 questions and is divided in four domains: inconvenience, restrictions, fears, and impact on daily life (9, 8, 8, and 5 questions, respectively).
  Each answer has five quantified items on a five category ordinal Likert scale with values ranging from 0 (no impact) to 4 (greatest negative impact). The average for each domain is calculated and used to obtain the final SIUP score (average of all domains, range from 0 to 4, 4 being the greatest negative impact).
  The second section, GQoL, has nine questions, also with a five-category ordinal Likert scale. It ranges from Very badly to Very well, with values ranging from -2 to +2, respectively.
  Final general QoL value is calculated as the average for the nine questions, also ranging from -2 to +2.
Short Form Qualiveen (SF-Qualiveen) | 6 months
  The SF-Qualiveen is a validated short version of the Qualiveen questionnaire and evaluates urinary-specific quality of life. The SF-Qualiveen consists of eight questions and reports on four domains of two questions each: bother with limitations, fears, feelings, and frequency of limitations. Responses are given on a 5-point Likert like scale, where a score of 0 indicates "no impact" and 4 "high impact." The SF-Qualiveen total score is calculated as the mean of the eight responses and the domain scores are calculated as the mean score of the responses per domain.
The King's Health Questionnaire (KHQ) | 6 months
  The King's Health Questionnaire (KHQ) is one of the most widely used for assessing QOL in patients with urinary incontinence (UI).The KHQ consists of two parts and 32 items. The first part (21 items) contains two single-item questions that address General Health Perception and Incontinence Impact and the following seven multi-item domains: Role, Physical, and Social Limitations, Limitations in Personal Relationship, Emotional Problems, Sleep and Energy Disturbances associated with UI, and Severity Measures for UI. The second part has an 11-item Symptom Severity Scale (SSS) that assesses the presence and severity of urinary symptoms. While the entire SSS is scored from 0 (best) to 30 (worst), the minimum possible score is 0 (best health) and the maximum possible score is 100 (worst health) for all other KHQ domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology Jagiellonian University, Krakow, Malopolska, Poland

REFERENCES:
- [Derived] Przydacz M, Kornelak P, Golabek T, Dudek P, Chlosta P. Polish versions of the Qualiveen and the SF-Qualiveen: Translation and validation of urinary disorder-specific instruments in patients with multiple sclerosis. Neurourol Urodyn. 2020 Aug;39(6):1764-1770. doi: 10.1002/nau.24419. Epub 2020 Jun 16. PMID 32542853